CLINICAL TRIAL: NCT06178588
Title: A Phase II Open-Label Study of Sacituzumab Govitecan in Patients With Previously Treated Locally Advanced, Recurrent, or Metastatic Cholangiocarcinoma
Brief Title: Sacituzumab Govitecan for the Treatment for Patients With Locally Advanced, Recurrent, or Metastatic Cholangiocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Anup Kasi, Principal Investigator, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00150700; NCI-2023-09080 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IIT-2023-SIGNA; STUDY00150700 (Other: University of Kansas Cancer Center); P30CA168524 (NIH)
Record Dates: First submitted 2023-12-09; First posted 2023-12-21 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Locally Advanced Cholangiocarcinoma; Metastatic Cholangiocarcinoma; Recurrent Cholangiocarcinoma; Stage III Hilar Cholangiocarcinoma AJCC v8; Stage III Intrahepatic Cholangiocarcinoma AJCC v8; Stage IV Hilar Cholangiocarcinoma AJCC v8; Stage IV Intrahepatic Cholangiocarcinoma AJCC v8
MeSH Terms: conditions — Cholangiocarcinoma; Klatskin Tumor | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Sacituzumab govitecan) (Experimental): Patients receive sacituzumab govitecan IV over 1-3 hours on days 1 and 8 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo tumor biopsy, PET/CT or MRI scans, and blood sample collection throughout the study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Biological: Sacituzumab Govitecan

INTERVENTIONS:
Procedure: Biopsy — Undergo tumor biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo PET/CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Biological: Sacituzumab Govitecan — Given IV
  Other Names: hRS7-SN38 Antibody Drug Conjugate; IMMU-132; RS7-SN38; Sacituzumab Govitecan-hziy; Trodelvy

SUMMARY:
This phase II trial tests how well sacituzumab govitecan works in treating patients with cholangiocarcinoma that has spread to nearby tissue or lymph nodes (locally advanced), that has come back after a period of improvement (recurrent) or that has spread from where it first started (primary site) to other places in the body (metastatic). Sacituzumab govitecan is a monoclonal antibody, called hRS7, linked to a toxic agent, called SN-38. HRS7 is a form of targeted therapy because it attaches to specific molecules (receptors) on the surface of tumor cells, known as TROP2 receptors, and delivers SN-38 to kill them.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine anti-tumor activity by overall response rate (ORR).

SECONDARY OBJECTIVES:

I. To determine treatment safety based on toxicities participants who have received at least one dose of sacituzumab govitecan.

II. To determine anti-tumor activity by progression free survival (PFS). III. To determine anti-tumor activity by disease control rate (DCR). IV. To determine overall survival (OS).

EXPLORATORY OBJECTIVES:

I. To determine if treatment will result in reduction of the circulating tumor deoxyribonucleic acid (DNA) as a measure of therapeutic response.

II. To determine relationship between tumor mutational profile (already performed as standard of care next generation sequencing [NGS] based test) to response.

OUTLINE:

Patients receive sacituzumab govitecan intravenously (IV) over 1-3 hours on days 1 and 8 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo tumor biopsy, positron emission tomography (PET)/computed tomography (CT) or magnetic resonance imaging (MRI) scans, and blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 30 days, and every 3 months for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Ability of participant or legally authorized representative (LAR) to understand this study, and participant or LAR willingness to sign a written informed consent
* Males and females age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days before day 1 of study treatment
* Locally advanced, recurrent or metastatic cholangiocarcinoma) after progressing or intolerant to at least one line of systemic therapy
* Adequate archival tissue from prior biopsy for biomarker evaluation or willingness to undergo tissue biopsy before treatment starts and on treatment. Patients who, in the opinion of the investigator, do not have tissue that can be safely biopsied are exempted
* Absolute neutrophil count ≥ 1.5 K/UL
* Hemoglobin ≥ 9 g/dL
* Platelets ≥ 100K/UL
* Creatinine clearance ≥ 30 mL/min as assessed by the Cockcroft-Gault equation {Cockcroft 1976} or Creatinine clearance ≥ 60 mL/min
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) OR direct bilirubin ≤ 1 x ULN
* Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 x ULN unless liver metastases are present, in which case they must be ≤ 5 x ULN
* Women of child-bearing potential and men with partners of child-bearing potential must agree to practice sexual abstinence or to use the forms of contraception for the duration of study participation and as follows:

  * Females: for 6 months following completion of therapy
  * Males: for 3 months following completion of therapy

Exclusion Criteria:

* Simultaneously enrolled in any therapeutic clinical trial
* Current or anticipating use of other anti-neoplastic or investigational agents while participating in this study
* Treatment with chemotherapy, biologics, or investigational agents that is not completed 4 weeks or 5 half-lives (whichever is longer) prior to first dose of study drug
* Diagnosed with a psychiatric illness or is in a social situation that would limit compliance with study requirements
* Other underlying medical condition that, in the opinion of the investigator, would impair the ability of the participant to receive or tolerate the planned treatment and follow-up; any known psychiatric or substance abuse disorders that would interfere with cooperating with the requirements of the study
* Is pregnant or breastfeeding
* Known homozygosity in the UGT1A1*28 allele associated with irinotecan toxicity
* Known hypersensitivity (≥ grade 3) to the study drug, its metabolites, or formulation excipient
* Requirement for ongoing therapy with (or prior use within 2 weeks of cycle 1, day 1) high dose systemic corticosteroids (≥ 20 mg of prednisone or its equivalent)
* Requirement for ongoing therapy with or prior use of UGT1A1 inhibitors/inducers
* Active grade 3 (per the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE], version 5.0) or higher viral, bacterial, or fungal infection within 2 weeks prior to the first dose of study treatment
* Have not recovered (i.e., ≥ grade 2 is considered not recovered) from adverse events (AEs) due to a previously administered agent.

  * Note: patients with any grade neuropathy or alopecia are an exception to this criterion and will qualify for the study.
  * Note: if patients received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Active central nervous system (CNS) metastases. Patients with treated CNS metastases are permitted on study if all the following are true:

  * CNS metastases have been clinically stable for at least 6 weeks prior to screening and baseline scans show no evidence of new or enlarged metastasis.
  * If requiring steroid treatment for CNS metastases, the patient is on a stable dose <10 mg/day of prednisone or equivalent for at least 2 weeks.
  * Patient does not have leptomeningeal disease
* Met any of the following criteria for cardiac disease:

  * Myocardial infarction or unstable angina pectoris within 6 months of enrollment.
  * History of serious ventricular arrhythmia (ie, ventricular tachycardia or ventricular fibrillation), high-grade atrioventricular block, or other cardiac arrhythmias requiring antiarrhythmic medications (except for atrial fibrillation that is well controlled with antiarrhythmic medication); history of QT interval prolongation.
  * New York Heart Association (NYHA) class III or greater congestive heart failure or left ventricular ejection fraction of < 40%
* Prior treatment with topoisomerase 1 inhibitors
* Have an active concurrent malignancy or malignancy within 3 years of study enrollment. Note: patients with a history of malignancy that have been completely treated, with no evidence of active cancer for 3 years prior to enrollment, or patients with surgically cured tumors with low risk of recurrence (e.g., nonmelanoma skin cancer, histologically confirmed complete excision of carcinoma in situ, or similar such as adequately treated basal or squamous cell carcinoma, non-melanomatous skin cancer, or curatively resected cervical cancer) are allowed to enroll
* Have active chronic inflammatory bowel disease (ulcerative colitis, Crohn's disease) or gastrointestinal (GI) perforation within 6 months of enrollment
* Currently receiving systemic antimicrobial treatment for active infection (viral, bacterial, or fungal) at the time of first dose of sacituzumab govitecan. Routine antimicrobial prophylaxis is permitted
* Have known history of human immunodeficiency virus (HIV)-1 or 2 (or positive HIV-1/2 antibody, if done at screening) with detectable viral load
* Have active hepatitis B virus (HBV) or hepatitis C virus (HCV). In patients with a history of HBV or HCV, patients with detectable viral loads will be excluded.

  * Patients who test positive for hepatitis B surface antigen (HBsAg). Patients who test positive for hepatitis B core antibody (anti-HBc) will require HBV DNA by quantitative polymerase chain reaction (PCR) for confirmation of active disease.
  * Patients who test positive for HCV antibody. Patients who test positive for HCV antibody will require HCV ribonucleic acid (RNA) by quantitative PCR for confirmation of active disease. Patients with a known history of HCV or a positive HCV antibody test will not require a HCV antibody at screening and will only require HCV RNA by quantitative PCR for confirmation of active disease
* Patients with active tuberculosis based on medical history
* Documented history of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction, or cardiac symptoms (including congestive heart failure) consistent with NYHA Class III-IV within 6 months prior to the first dose of sacituzumab govitecan
* Radiotherapy or major surgery within 2 weeks prior to first dose of study drug. Patient must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment
* Administration of a live, attenuated vaccine within 30 days prior to first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, BCG, and typhoid vaccine.

  * Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist [registered trademark]) are live attenuated vaccines and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | From start of treatment, up to 2 years
  Defined as best response recorded from the start of the treatment until the end of treatment (taking into account any requirement for confirmation).
  Measured by computed tomography (CT) (magnetic resonance imaging [MRI] if CT contraindicated) Response Evaluation Criteria in Solid Tumors (RECIST 1.1). Will be reported as a proportion with corresponding 90% confidence interval.

SECONDARY OUTCOMES:
Incidence of adverse events | From enrollment to 30 days after last administration of study treatment
  Measured by Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0.
Anti-tumor activity: Duration of response | From enrollment to end of follow up, up to 2 years
  Measured by RECIST 1.1
Anti-tumor activity: Disease control rate | From enrollment to end of follow up, up to 2 years
  Measured by RECIST 1.1
Progression free survival | From start of treatment until objective tumor progression or death, up to 2 years
  Measured by survival curve and the medical record. Will be reported using Kaplan Meier estimates of the median along with a 90% confidence interval.
Overall survival | From start of treatment to death, up to 2 years
  Measured by survival curve and the medical record. Will be reported using Kaplan Meier estimates of the median along with a 90% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Anup K Kasi Loknath Kumar, Principal Investigator — University of Kansas
Locations (1):
- University of Kansas Cancer Center, Kansas City, Kansas, United States